CLINICAL TRIAL: NCT00225043
Title: A Randomized, Double-Blind, Trial Comparing Epinephrine Versus Phenylephrine as a Vasoconstrictor in Regional Anesthesia for Upper Extremity Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Presbyterian Brooklyn Methodist Hospital (Other)
Responsible Party: Joel Yarmush, New York Methodist Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 299
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2008-06-02 (Estimated); Status verified 2008-05

CONDITIONS: Healthy
MeSH Terms: interventions — Epinephrine; Phenylephrine

INTERVENTIONS:
Drug: Epinephrine/phenylephrine

SUMMARY:
The study involves research, the purpose of which is to compare three different drug mixtures (Epinephrine, Phenylephrine 25 µg, or Phenylephrine 50 µg). Specifically, how long each medicine lasts will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder surgery with regional anesthesia

Exclusion Criteria:

* Shoulder surgery with general anesthesia unhealthy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Yarmush, MD, MPA, Principal Investigator — New York Presbyterian Brooklyn Methodist Hospital
Locations (1):
- New York Methodist Hospital, Brooklyn, New York, United States